CLINICAL TRIAL: NCT00700700
Title: Effects of Cardiac Resynchronization Therapy on Dyspnea and Exercise Tolerance in Patients With Congestive Heart Failure
Brief Title: Cardiac Resynchronization Therapy, Dyspnea and Exercise Tolerance in Patients With Congestive Heart Failure (CHF)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped due to an inability to recruit eligible subjects.
Sponsor: Queen's University (Other)
Responsible Party: Dr. Chris M. Parker, Assistant Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMED-1082-07
Record Dates: First submitted 2008-05-16; First posted 2008-06-19 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Cardiac Resynchronization Therapy; Dyspnea; Exercise Tolerance
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRT-ON/CRT-OFF (Active Comparator): Group initially randomized to CRT-ON, then cross-over to CRT-OFF
  Interventions: Device: Active Cardiac Resynchronization Therapy (CRT)
- CRT-OFF/CRT-ON (Active Comparator): Group initially randomized to CRT-OFF, then cross-over to CRT-ON
  Interventions: Device: Active Cardiac Resynchronization Therapy (CRT)

INTERVENTIONS:
Device: Active Cardiac Resynchronization Therapy (CRT) — Initiation of active biventricular pacing/cardiac resynchronization therapy
  Devices by Medtronic:
  1. Insync Sentry 7298 & 7299
  2. Concerto C174 ASK (Most frequently implanted)
  3. Insync III 8042 (PM)
  Devices by Guidant/Boston Scientific:
  1. Contak Renewal 4 H190 & H199
  2. Contak Renewal 3 H127
  Devices by ELA/Sorin:
  1. Ovatio CRT 6750
  Other Names: Received one of the above devices used in 2007-2008 at Kingston General Hospital.

SUMMARY:
A new therapy for patients with advanced heart failure (HF) involves the implantation of a specialized pacemaker device (Cardiac Resynchronization Therapy, CRT) that attempts to restore the synchronized contraction of the ventricular chambers of the heart. In some people, CRT improves exertional breathlessness and allows them to exercise for longer periods. However, to date, the mechanisms by which CRT improves symptoms and exercise tolerance is unknown. This study will use in-depth cardiopulmonary exercise testing and pulmonary function testing to explore these mechanisms in greater detail.

ELIGIBILITY:
Inclusion Criteria:

* clinically stable
* being considered for implantation of biventricular pacemaker for CRT
* LVEF <35%
* QRS duration >120 msec
* NYHA III-IV functional class
* optimized pharmacologic management of CHF
* no recent (<1 month) episodes of decompensated CHF

Exclusion Criteria:

* inability to perform cycle ergometry or comply with testing
* uncontrolled ischemic heart disease
* coronary revascularization within 3 months of study entry
* concurrent primary lung disease
* current use of ambulatory oxygen
* rhythm other than sinus
* dependency on pacemaker therapy as a consequence of bradyarrhythmias
* severe valvulopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Exercise endurance time | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chris M. Parker, MD, MSc, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada